CLINICAL TRIAL: NCT06856785
Title: Resonance Tube Voice Therapy Versus Smith Accent Therapy in The Management of Non-Organic Dysphonia in Adults
Brief Title: Management of Non-Organic Dysphonia in Adults.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shereen Mohamed Hamed, Phoniatric Resisdent Physician, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-2-02MS
Record Dates: First submitted 2025-02-23; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Functional Dysphonia; Resonance Tube Voice Therapy; Smith Accent Method Therapy
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-organic (Functional) dysphonia patients will receive Smith Accent Voice Therapy (No Intervention): The patient was advised to vocal hygiene and to correct the faulty vocal technique by a-diaphragmatic breathing in the sitting position by Using the newly acquired diaphragmatic breathing, the patient is allowed to "sing" the various vowels (/a/, /i/, and /u/), "the largo with one accentuation, the andante with three accentuations, and the fastest, allegro, with five accentuations". b-Body and arm movements during dynamic vowel exercises.
  Transfer and carry over to connected speech by (the gradual stage-wise transformation from vowel play to connected speech, repeating short phrases after the therapist, reading short phrases with pauses, monologue with short phrases with suitable pauses, dialogue, applying the same pattern)
- Non-organic (Functional) dysphonia patients will receive Resonance Tube Voice Therapy (Active Comparator): The patient sits comfortably with their back straight, holding the tube between their thumb and index fingers, maintaining 1 mm between their teeth, and ensuring no air leak between their lips and the tube. A 1-liter wide plastic container is used, filled with water, with the free end of the tube submerged 2 cm below the water's surface. The patient is instructed to take enough time to relax their respiratory muscles and phonate into the tube to create air bubbles on the water's surface, starting with monotonous words and progressing to different intonations. There are 2-minute rest periods between exercises, and the patient should drink water to prevent dryness. Sessions occur in the clinic until the patient can perform the exercises independently without effort, after which the pathologist may allow practice at home. The patient receives written instructions to practice 10 times daily for 2 minutes each, with 1 hour between practices for 6 weeks.
  Interventions: Other: Resonance Tube Voice Therapy in Water

INTERVENTIONS:
Other: Resonance Tube Voice Therapy in Water — Resonance Tube of 28 cm in length and 9 mm diameter for adults will be submerged into a bowl of water .Both flexible soft walled tubes,glass tubes or straws can be used
  Other Names: Smith Accent Voice Exercises
  Arms: Non-organic (Functional) dysphonia patients will receive Resonance Tube Voice Therapy

SUMMARY:
The purpose of this study is to determine the effect of a semi-occluded vocal tract training program, "Resonant Tube Therapy," versus the "Traditional Smith-accent Method" on the quality of voice in patients with Non-Organic "Functional" dysphonia.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with non-organic functional dysphonia with or without Minimally Associated Pathological lesions and referred for voice therapy. The diagnosis was based on the results of the routine clinical assessment of cases of voice disorders by a phoniatrician in the voice clinic.
* Patients 'ages between 15 - 60 years old.
* Native speakers of Arabic.
* Language comprehension adequate for the task.

Exclusion Criteria:

* Patients with organic voice disorders.
* Patients with aphonia or Phon asthenia.
* Females within the week of their menstrual cycle or menstruating at the time of data collection to control for the possible hormonal effects or premenstrual water retention on voice quality.
* History of severe respiratory allergies, thyroid pathologies, neuro-motor impairment, hearing impairment, psychiatric problems and physically limiting diseases that might interfere with study completion.
* Those on any regular medication that might affect voice quality.
* Speech disorders.
* Cigarette smoking, alcohol, or drug abuse for the past 5 years.
* Patients with previous micro laryngeal surgery.
* Patients with gastrointestinal reflux disease.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Voice quality improvement in functional (non-organic) dysphonia adult patients | 12 weeks following end of the treatment
  Patient evaluation will be conducted before and after the voice therapy sessions for the two groups by Voice Handicap Index (VHI).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No